CLINICAL TRIAL: NCT06496620
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Dose-Ranging Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Solrikitug in Participants With Chronic Obstructive Pulmonary Disease (ZION)
Brief Title: A Study to Evaluate Solrikitug in Participants With COPD (ZION)
Acronym: ZION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Uniquity One (UNI) (Industry)
Collaborators: DevPro Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSI-8226-205
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Biological: Solrikitug High Dose (Experimental): Solrikitug
  Interventions: Biological: Biological: Solrikitug high dose
- Placebo (Other): Placebo
  Interventions: Other: Placebo
- Biological: Solrikitug Low Dose (Experimental): Solrikitug
  Interventions: Biological: Biological: Solrikitug low dose

INTERVENTIONS:
Biological: Biological: Solrikitug low dose — Solrikitug subcutaneous injection
  Arms: Biological: Solrikitug Low Dose
Biological: Biological: Solrikitug high dose — Solrikitug subcutaneous injection
  Arms: Biological: Solrikitug High Dose
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
A Randomized, Double-blind, Placebo-controlled, Multiple Dose-Ranging Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Solrikitug in Participants with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
This is a 12-week randomized, double-blind, placebo-controlled clinical study to evaluate the safety, tolerability, PK, immunogenicity, and pharmacodynamics of 2 dose levels of solrikitug versus placebo on top of standard of care in participants with COPD.

Approximately 171 eligible participants with COPD will be randomized at approximately 60-90 sites. Participants will receive solrikitug, or placebo, administered via subcutaneous injection at the study site, over a 12-week treatment period. The study also includes a post-treatment follow-up period of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 40 years of age and no older than 75 years.
* Documented diagnosis of COPD for at least 12 months prior to Screening, defined by the GOLD Guidelines (2023), and elevated blood eosinophils at screening.
* At Screening FEV1/FVC ratio must be <0.70, and Post-bronchodilator FEV1 must be ≥40% to <80% predicted normal value calculated using Global Lung Function Initiative (GLI) reference equations (Cooper et al 2017).
* Symptomatic (COPD Assessment Test [CAT] Score ≥10) at Screening Visit 1.
* Participants must be on 2 or more inhaled maintenance medications for management of their COPD, for at least 3 months prior to screening.

Exclusion Criteria:

* Female participant who is pregnant or breastfeeding.
* Participant has a known hypersensitivity to any component of the formulation of solrikitug, including any of the excipients, or a history of anaphylactic reaction to any therapeutic monoclonal antibody.
* Participant has history or evidence of any clinically significant cardiovascular, hematologic, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy, or any other condition that in the opinion of the Investigator or Medical Monitor might obfuscate the study data.
* Any other pulmonary disease than COPD that in the opinion of the Investigator, the severity of the disorder would impact the conduct of the study.
* Undergone major lung surgery, within 1 year of Screening Visit 1.
* Participant has a lower respiratory tract infection that required antibiotics within 6 weeks prior to Screening.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in blood eosinophil counts | Through week 12
  To assess the effect of multiple doses of solrikitug on blood eosinophil counts compared with placebo

SECONDARY OUTCOMES:
Change from baseline in FEV1 Adverse events (AEs) and serious adverse events (SAEs) | Through week 12 To week 28
  To assess the safety and tolerability of multiple doses of solrikitug

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Lee, MD, Study Director — Vice President, Clinical Research
Locations (90):
- United States (87):
  - Research Site 034, Birmingham, Alabama
  - Research Site 099, Peoria, Arizona
  - Research Site 051, Sun City, Arizona
  - Research Site 033, Tempe, Arizona
  - Research Site 095, Tucson, Arizona
  - Research Site 031, Lancaster, California
  - Research Site 107, Long Beach, California
  - Research Site 032, Los Angeles, California
  - Research Site 018, Newport Beach, California
  - Research Site 041, Oxnard, California
  - Research Site 056, Rancho Cucamonga, California
  - Research Site 020, Englewood, Colorado
  - Research Site 070, Brooksville, Florida
  - Research Site 049, Clearwater, Florida
  - Research Site 002, Clearwater, Florida
  - Research Site 035, Cutler Bay, Florida
  - Research Site 077, DeLand, Florida
  - Research Site 064, Hialeah, Florida
  - Research Site 057, Homestead, Florida
  - Research Site 111, Miami, Florida
  - Research Site 101, Miami, Florida
  - Research Site 059, Miami, Florida
  - Research Site 098, Miami, Florida
  - Research Site 004, Miami, Florida
  - Research Site 038, Miami Gardens, Florida
  - Research Site 055, Miami Lakes, Florida
  - Research Site 013, Orlando, Florida
  - Research Site 007, Sarasota, Florida
  - Research Site 067, Tamarac, Florida
  - Research Site 001, Tampa, Florida
  - Research Site 108, Adairsville, Georgia
  - Research Site 046, Dublin, Georgia
  - Research Site 110, East Point, Georgia
  - Research Site 003, Rincon, Georgia
  - Research Site 021, Meridian, Idaho
  - Research Site 079, Peoria, Illinois
  - Research Site 022, Merrillville, Indiana
  - Research Site 042, Lexington, Kentucky
  - Research Site 026, Metairie, Louisiana
  - Research Site 097, Shreveport, Louisiana
  - Research Site 017, South Dartmouth, Massachusetts
  - Research Site 114, Dearborn, Michigan
  - Research Site 037, Farmington Hills, Michigan
  - Research Site 085, Southfield, Michigan
  - Research Site 009, Saint Charles, Missouri
  - Research Site 062, Missoula, Montana
  - Research Site 015, Henderson, Nevada
  - Research 044, Cortland, New York
  - Research Site 044, Cortland, New York
  - Research Site 043, Horseheads, New York
  - Research Site 050, Charlotte, North Carolina
  - Research Site 005, Gastonia, North Carolina
  - Research Site 104, Greensboro, North Carolina
  - Research Site 008, High Point, North Carolina
  - Research Site 039, Huntersville, North Carolina
  - Research Site 006, Wilmington, North Carolina
  - Research Site 014, Winston-Salem, North Carolina
  - Research Site 036, Columbus, Ohio
  - Research Site 086, Lima, Ohio
  - Research Site 115, Edmond, Oklahoma
  - Research Site 047, Grants Pass, Oregon
  - Research Site 011, Medford, Oregon
  - Research Site 083, DuBois, Pennsylvania
  - Research Site 053, Pittsburgh, Pennsylvania
  - Research Site 023, Anderson, South Carolina
  - Research Site 028, Columbia, South Carolina
  - Research Site 030, Gaffney, South Carolina
  - Research Site 027, Greenville, South Carolina
  - Research Site 010, Rock Hill, South Carolina
  - Research Site 024, Spartanburg, South Carolina
  - Research Site 029, Union, South Carolina
  - Research Site 040, Hendersonville, Tennessee
  - Research Site 048, Knoxville, Tennessee
  - Research Site 016, Boerne, Texas
  - Research Site 076, Brownsville, Texas
  - Research Site 112, Carrollton, Texas
  - Research Site 012, Dallas, Texas
  - Research Site 089, Greenville, Texas
  - Research Site 051, Houston, Texas
  - Research Site 060, Houston, Texas
  - Research Site 025, Houston, Texas
  - Research Site 087, Katy, Texas
  - Research Site 012, McKinney, Texas
  - Research Site 084, Mesquite, Texas
  - Research Site 109, Splendora, Texas
  - Research Site 088, Layton, Utah
  - Research Site 019, Hampton, Virginia
- Research Site 090, Tarragindi, Queensland, Australia
- Research Site 094, Waikanae, New Zealand
- Research Site 096, High Wycombe, United Kingdom